CLINICAL TRIAL: NCT05123872
Title: GleichStrom UND Depression: Anwendung zu Hause Ohne Anreise Zur Medbo (Transcranial Direct Current Stimulation and Depression: Home Treatment)
Brief Title: Transcranial Direct Current Stimulation as Home Treatment in Depression
Acronym: GSUND_DAHOAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Collaborators: neurocare group AG (Unknown)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Clinical Professor, MD, Ph.D., University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-2091-101
Record Dates: First submitted 2021-09-21; First posted 2021-11-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prefrontal tDCS at home (Experimental): trancranial direct current stimulation 30 sessions within 6 weeks (treatment on working days) 2mA with cathode on the right and anode an the left side
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — trancranial direct current stimulation 30 sessions within 6 weeks (treatment on working days) 2mA with cathode on the right and anode an the left side

SUMMARY:
In this one-armed study the feasibility and effectiveness of a home treatment with transcranial direct currect stimulation in depression will be investigated.

DETAILED DESCRIPTION:
In this one-armed study at least 10 patients with depression will be included who will get treatment with transcranial direct currect stimulation at home. One visit in the hospital before and one visit after the treatment are necessary. The correct application of the device by the patients will be ensured by video counseling and monitoring. Treatment will last six weeks with 2 mA applied every working day for 20min with prefrontal montage.

Aim of the study is the evaluation of the feasibility of this home treatment (usability of the device, compliance of patients, usability of the video contacts), the effectiveness (clinical ratings) and the tolerability of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* depressive episode according to ICD-10
* moderate depression according to clinical impression or Hamilton depression rating scale
* gender: all sexes
* age: 18-70 years
* stable medication if possible
* no or stable treatment of depression
* residence in Germany and mother language German
* written informed consent

Exclusion Criteria:

* contraindications for transcranial direct current stimulation
* neurological conditions
* participiation in another study
* pregnancy and lactation period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Usability for the patients | 6 weeks
  Rating of the usability of the treatment (home treatment and video monitoring) with the user experience questionnaire [1-7, 26 items, the higher the better] and open feedback
Usability for the handlers/clinicians | 6 weeks
  Rating of the usability of the treatment (home treatment and video monitoring) with the user experience questionnaire [1-7, 26 items, the higher the better] and open feedback
Compliance 1 (Number of days out of 30 the patients used the device) | 6 weeks
  Number of days out of 30 the patients used the device
Compliance 2 (Number of patients who completed the treatment regulary) | 6 weeks
  Number of patients who completed the treatment regulary
Efficiancy 1 (Number of responders according the the clinical global impression change score for patients in the per protocol analysis) | 6 weeks
  Number of responders according the the clinical global impression change score for patients in the per protocol analysis
Efficiancy 2 (Effect size for change of depressivity for patients in the per protocol analysis measured with the Hamilton depression rating scale (21 items)) | 6 weeks
  Effect size for change of depressivity for patients in the per protocol analysis measured with the Hamilton depression rating scale (21 items)
Stability of effects 1 (Number of responders according the the clinical global impression change score) | 18 weeks
  Number of responders according the the clinical global impression change score
Stability of effects 2 (Effect size for change of depressivity for patients in the per protocol analysis measured with the Hamilton depression rating scale (21 items)) | 18 weeks
  Effect size for change of depressivity for patients in the per protocol analysis measured with the Hamilton depression rating scale (21 items)

SECONDARY OUTCOMES:
Hamilton depression rating scale | 18 weeks
  Depression rating scale (0-65, the lower the better)
Major Depression Inventory | 18 weeks
  Depression inventory (0-50, the lower the better)
WHO Quality of life scale (abbreviated Version) (WHOQOL-BREF) | 18 weeks
  Quality of life scale inventory (4-20, the higher the better)
Clincial Global Impression change | 18 weeks
  Clincial Global Impression (1-7, the lower the better)
Pittsburgh sleep quality index | 18 weeks
  sleep inventory (0-21, the lower the better)
Depression anxiety stress scale (DASS) | 18 weeks
  Depression, anxiety and stress inventory (each 0-21, the lower the better)
Personality styles and disorder inventory | 18 weeks
  Depedence of treatment effect from personality as measured with the Personality styles and disorder inventory (PSDI) (T-value norms, values around 50 are normal)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, PhD, Principal Investigator — University of Regensburg
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No